CLINICAL TRIAL: NCT02760134
Title: The Influence of Super-Mini Percutaneous Nephrolithotomy on Renal Pelvic Pressure In Vivo
Brief Title: The Influence of SMP on Renal Pelvic Pressure In Vivo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Guohua Zeng, Vice President of the Hospital, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MRER(14)2016
Record Dates: First submitted 2016-04-30; First posted 2016-05-03 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Renal Calculi
Keywords: Super-Mini Percutaneous Nephrolithotomy(SMP); Renal Pelvic Pressure
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMP with F14 sheath (Other): Patients undergo Super-Mini Percutaneous Nephrolithotomy with F14 suction-evacuation sheath.
  Interventions: Procedure: Super-Mini Percutaneous Nephrolithotomy
- SMP with F12 sheath (Other): Patients undergo Super-Mini Percutaneous Nephrolithotomy with F12 suction-evacuation sheath.
  Interventions: Procedure: Super-Mini Percutaneous Nephrolithotomy

INTERVENTIONS:
Procedure: Super-Mini Percutaneous Nephrolithotomy — Patients undergo Super-Mini Percutaneous Nephrolithotomy

SUMMARY:
Percutaneous nephrolithotomy (PCNL) is a well-established treatment modality for renal stones. It offers a high stone free rates and less invasive than open surgery. Nevertheless PCNL is an invasive and technically demanding procedure with inherent risks and complications. The most troublesome morbidities are bleeding and injury to the kidney and its adjacent structures. Complications of PCNL tend to be associated with the accuracy of tract placement and the size of the nephrostomy tract. To improve the safety of PCNL, there is a trend toward using smaller and smaller nephrostomy tracts . With the smaller nephrostomy tract, there also arise the problems of compromised visual field and increased difficulty in stone extraction. Increase irrigation using pressure pump might improve the visualization and the passive egress of the stone fragments, but it also may concomitantly increase the intra-luminal pressure.

The present system of Super-Mini percutaneous nephrolithotomy (SMP) was developed to address many of these deficiencies. The basic components of SMP system are an 8.0 F miniaturized nephroscope with a newly designed irrigation-suction sheath with enhanced irrigation capability and modified nephrostomy sheath with continuous negative pressure aspiration. Its design was intended not only to prevent the excessive intrarenal pressure but also improve the visualization and the stone fragments extraction.

Little was known about renal pelvic pressure in vivo during SMP and about any correlation it might have had with postoperative fever and urosepsis. We measure the renal pelvic pressure during SMP to determine whether it will improve the renal pelvic pressure and improve the incidence of postoperative fever.

DETAILED DESCRIPTION:
To evaluate the influence of SMP on renal pelvic pressure for the treatment of renal calculi measuring smaller than 25 mm. Investigators will do a single center randomized open-label trial，and investigators plan to perform this study in the First Affiliated Hospital of Guangzhou Medical University of China.

Investigators plan to beginning their study at April in 2016 and end at March in 2018.One hundred patients with renal calculi measuring smaller than 25 mm will be enrolled in this study. By simple random sampling technique, patients will be assigned to two 50-patient groups(group 1:F14,group2 :F12).All the patients will be diagnosed definitely before operations with non-contrast CT. Patients with positive preoperative urine culture should be treated with suitable antibiotics based on the culture sensitivity result for at least 72h before SMP. Patients who have negative urine culture should receive a single dose of broad spectrum antibiotic prophylaxis just prior to the procedure.

Surgical technique Routine preoperative preparations are carried out as for conventional percutaneous surgery. Under general anesthesia and with the patient in the lithotomy position, an open-ended 5F ureteral catheter is advanced into the renal pelvis under direct vision. The patient is then turned into the prone position. Percutaneous access is achieved using an 18-gauge coaxial needle to puncture the selected calyx under fluoroscopic or ultrasonic guidance. The success of the puncture is confirmed both by the free flow of the irrigation fluid and by fluoroscopic images. Using a guidewire, the dilatation is carried out with 10 F fascial dilators. Thenan irrigation-suction straight sheath, with the obturator, is advanced over the guidewire and introduced into the pelvicalyceal system. The guidewireis then removed, and the "handle" is connected to the straight sheath. The irrigation port of the irrigation-suction sheath is connected to an irrigation pump. The oblique tube of the sheath is connected to the specimen collection bottle, and the bottle then to the negative pressure aspirator. The irrigation fluid pressure is set as 200-250 mmHg. The suction pressure is controlled to a setting of 100-150 mmHg. The irrigation is delivered through the irrigation channel of the sheath. Thus, a one-way flow is created as the inflow that comes out of the irrigation channel of the sheath is immediately aspirated through the suction conduitof the sheath. Stone fragmentation is accomplished using either holmium laser or pneumatic lithotripter. The tiny pulverized stone fragments will pass around the scope and evacuate through the oblique sluice. If the stone fragments are too large to pass around the scope inside the sheath, the scope can be withdrawn slowly to proximal to the bifurcation in order to create an unobstructed channel for larger fragments evacuation. At the end of the procedure, a single fluoroscopic image is obtained to assess the stone-free status. A Double-J stent is placed only when there is the presence of an obstructing inflammatory ureteric edema, ureteropelvic junction obstruction, or concurrent treatment of ipsilateral ureteric stone with rigid ureteroscope. The sheath is removed, and the wound is either sutured or seal with absorbable gelatin. For patients with significant bleeding or extravasation, a nephrostomy tube is placed.

Measurement of Renal Pelvic Pressure In Vivo While preparing for the SMP, the open-ended ureteric catheter, which had been inserted into the renal collecting system retrogradely, was connected to the invasive blood pressure channel of patient monitor with a baroceptor. The baroceptor was fixed onto the horizontal plane of renal pelvis; after a zero adjustment, the measurement of renal pelvic pressure was in session. A computer collected the renal pelvic pressure data each second. Any factor that caused a high renal pelvic pressure was noticed .

Data collection Data for the 2 groups -demographic characteristics, site of access ,Hb decrease, CRP increase, WBC increase, postoperative pain, operation time, hospital stay, cases of tubeless, postoperative infection complications (systemic inflammatory response syndrome, urosepsis), stone clearance rate and the need for auxiliary treatment are compared.

Primary study endpoint: The renal pelvic pressure. Secondary endpoint: Postoperative systemic inflammatory response syndrome or urosepsis, stone clearance rate, operation time, hospital stay.

Demographic characteristics include age, sex, BMI, stone size and location, etc.

Stone size is defined as the maximum diameter. Operation time is recorded from the time of the first percutaneous renal puncture to the completion of the stone removal.

Hospital stay are rounded to the nearest whole day and calculated from the day of surgery to the day of discharge.

Postoperative pain (visual analogue scale [VAS], use of analgesics) and Postoperative comfort scores (Bruggrmann comfort scale [BCS]) will be recorded.

The rate of hemoglobin decrease is assessed by comparing the preoperative Hb level with 24-hour postoperative Hb level.

Primary SFR and final SFR is assessed by KUB at day 1 and 1 month after operation.

Stone-free status are defined as either the absence of any residual stone fragments or the presence of clinically insignificant residual stone fragments in the kidney which were defined as ≦ 3mm, asymptomatic, non-obstructive and non-infectious stone particles.

If the procedure is considered as successful, the double J stent is removed as outpatient after 2 weeks. Follow-up including KUB or non-contrast CT will be generally scheduled in 1 month.

Bleeding severity is judged by the treating physician, and transfusions are administered according to local practice guideline.

Complications of all patients are recorded according to modified Clavien classification system.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 70 years
2. Anesthesia rating(ASA) score 1 and 2
3. No obvious preoperative symptoms of infection(chills, fever, etc.)
4. Symptomatic renal calculi and diameter smaller than 25mm

Exclusion Criteria:

1. Couldn't tolerate SMP
2. Hydronephrosis
3. Ureteral calculi or urinary tract anomalies, stricture or obstruction
4. Abdominal cavity effusion affecting breathe
5. Patients with congenital anomalies, e.g. ectopic kidney, polycystic
6. Patients who underwent transplant or urinary diversion
7. Uncorrected coagulopathy
8. Patient undergoing any other surgical procedure during the same admission. (e.g. ureteroscopy)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
The renal pelvic pressure | Every one second intraoperatively
  The measurement of renal pelvic pressure was collected each second by the computer.

SECONDARY OUTCOMES:
Postoperative systemic inflammatory response syndrome | Within 1 month postoperatively
  Postoperatively patients were monitored for signs of SIRS, which is manifested by two or more of the following conditions: (1)Temperature > 38°C or < 36°C,(2) Heart rate > 90 bpm,(3) Respiratory rate > 20 breaths/min or PaCO2 < 32 mmHg (< 4.3 kPa),(4) WBC > 12,000 cells/mm3 or < 4,000 cells/mm3 or > 10% immature (band) forms.
Operation time | Intraoperatively
  Operation time is the duration of the operation from the time of the first percutaneous renal puncture to the completion of the stone removal.
Hospital stay | Within 1 month postoperatively
  Hospital stay is rounded to the nearest whole day and calculated from the day of surgery to the day of discharge.
Hemoglobin decrease | Within 24 hours after the operation
  The rate of hemoglobin decrease is assessed by comparing the preoperative Hb level with 24-hour postoperative Hb level.
Stone-free status | Within 1 month postoperatively
  Stone-free status are defined as either the absence of any residual stone fragments or the presence of clinically insignificant residual stone fragments in the kidney which were defined as ≦ 3mm, asymptomatic, non-obstructive and non-infectious stone particles.

CONTACTS AND LOCATIONS:
Overall Officials: Guohua Zeng, PH.D and M.D, Study Chair — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- epartment of Urology, Minimally Invasive Surgery Center, The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China